CLINICAL TRIAL: NCT04598789
Title: Study to Evaluate the Outcome of HSCT Mismatch Unrelated Donors
Brief Title: A Multicentre, Retrospective Study to Evaluate the Outcome of HSCT Mismatch Unrelated Donors
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Director, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: Allo MM HSCT
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Leukemia, Myeloid
MeSH Terms: conditions — Leukemia, Myeloid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention, observational study

SUMMARY:
The primary endpoint of the study was the acute GvHD incidence, the secondary endpoints were chronic GvHD incidence, overall survival (OS), transplant related mortality (TRM) incidence, relapse incidence (RI) and neutrophil and platelets engraftment after GvHD prophylaxis with ATG-CSA-MTX or PTCy-MMF-FK506

ELIGIBILITY:
Inclusion Criteria:

* children and adults)
* HSCT from a one-antigen mismatch unrelated donors
* Treated at the Centro Trapianti Metropolitano di Torino between 2012 to 2017

Exclusion Criteria: none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (children and adults) having HSCT from a one-antigen mismatch unrelated donors and treated at the Centro Trapianti Metropolitano di Torino between 2012 to 2017
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
acute GvHD incidence | 2012-2017

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Turin, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Berger M, Barone M, Spadea M, Saglio F, Pessolano R, Fagioli F. HSCT with mismatched unrelated donors: Bone marrow versus peripheral blood stem cells sources in pediatric patients. Pediatr Transplant. 2022 Jun;26(4):e14233. doi: 10.1111/petr.14233. Epub 2022 Jan 28. PMID 35092128